CLINICAL TRIAL: NCT02696954
Title: A Randomized, Open-Label Study to Evaluate Potential Pharmacokinetic Interactions of Orally Administered Artemether-lumefantrine, Amodiaquine and Primaquine in Healthy Adult Subjects
Brief Title: Study of Artemether-lumefantrine, Amodiaquine and Primaquine in Healthy Subjects
Acronym: ALAQPQ
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other); Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALAQPQ
Record Dates: First submitted 2016-02-18; First posted 2016-03-02 (Estimated); Last update posted 2019-06-28 (Actual); Status verified 2019-05

CONDITIONS: Pharmacokinetic; Drug Combination; Healthy
Keywords: Artemether-lumefantrine; Amodiaquine; Primaquine
MeSH Terms: interventions — Artemether, Lumefantrine Drug Combination; Amodiaquine; Primaquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental)
  Interventions: Drug: Artemether-lumefantrine; Drug: Amodiaquine; Drug: Artemether-lumefantrine + Amodiaquine; Drug: Primaquine; Drug: Artemether-lumefantrine + Primaquine; Drug: Artemether-lumefantrine + Amodiaquine + Primaquine
- Group B (Experimental)
  Interventions: Drug: Amodiaquine; Drug: Artemether-lumefantrine; Drug: Artemether-lumefantrine + Amodiaquine; Drug: Primaquine; Drug: Artemether-lumefantrine + Amodiaquine + Primaquine; Drug: Artemether-lumefantrine + Primaquine

INTERVENTIONS:
Drug: Artemether-lumefantrine — Artemether-lumefantrine on Day 0, 1 and 2 Washout period: more than 6 weeks
  Arms: Group A
Drug: Amodiaquine — Amodiaquine on Day 0, 1 and 2 Washout period: more than 6 weeks
Drug: Artemether-lumefantrine — Artemether-lumefantrine on Day 0, 1 and 2 Washout period: more than 6 weeks
  Arms: Group B
Drug: Artemether-lumefantrine + Amodiaquine — Artemether-lumefantrine + Amodiaquine on Day 0, 1 and 2 Washout period: more than 6 weeks
Drug: Primaquine — Primaquine on Day 0 Washout period: more than 1 week
Drug: Artemether-lumefantrine + Primaquine — Artemether-lumefantrine on Day 0, 1 and 2 + Primaquine on Day 0 Washout period: more than 6 weeks
  Arms: Group A
Drug: Artemether-lumefantrine + Amodiaquine + Primaquine — Artemether-lumefantrine Day 0, 1 and 2 + Amodiaquine on Day 0, 1 and 2 + Primaquine on Day 0 Washout period: more than 6 weeks
Drug: Artemether-lumefantrine + Primaquine — Artemether-lumefantrine on Day 0, 1 and 2 + Primaquine on Day 0
  Arms: Group B

SUMMARY:
Primary Objective

* To characterize the potential pharmacokinetic interactions of artemether -lumefantrine, amodiaquine and primaquine in healthy adult subjects.

Secondary Objectives

* To characterize the pharmacokinetic properties of artemether-lumefantrine, amodiaquine and primaquine when given alone and in combination.
* To evaluate the safety and tolerability of co-administered artemether-lumefantrine, amodiaquine and primaquine.
* To investigate pharmacogenetic polymorphisms affecting drug levels of artemether-lumefantrine, amodiaquine and primaquine and their metabolites.

DETAILED DESCRIPTION:
The study design is an open-label pharmacokinetic study in healthy G6PD normal Thai subjects. This study will enroll 16 healthy subjects. Participants who pass the screening process will have 6 admissions in the hospital to receive 6 drug regimens as below

First admission visit: The subject may be randomized to receive either Artemether-Lumefantrine or Amodiaquine with more than 6 weeks washout period before second admission visit.

Second admission visit: Subject who receives Artemether-Lumefantrine from previous visit will receive amodiaquine in this visit and vice versa. This visit will required more than 6 weeks washout period before third admission visit.

Third admission visit: Every subject will receive Artemether-lumefantrine and Amodiaquine with more than 6 weeks washout period before forth admission visit.

Forth admission visit: Every subject will receive Primaquine with more than 1 week washout period before fifth admission visit.

Fifth admission visit: Subject may randomize to receive either Artemether-Lumefantrine and Primaquine or Artemether-Lumefantrine and Amodiaquine and Primaquine in this visit with more than 6 weeks washout period before sixth admission visit.

Sixth admission visit: Subject who receives Artemether-Lumefantrine and Amodiaquine and primaquine from previous visit will receive Artemether-Lumefantrine and Primaquine in this visit and vice versa.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy as judged by a responsible physician with no abnormality identified on a medical evaluation including medical history and physical examination.
2. Male or female non-smoker aged between 18 years to 60 years.
3. A female is eligible to enter and participate in this study if she is:

   * of non-childbearing potential including pre-menopausal females with documented (medical report verification) hysterectomy or double oophorectomy
   * or postmenopausal defined as 12 months of spontaneous amenorrhea or 6 months of spontaneous amenorrhea with serum follicle stimulating hormone levels >40 mIU/mL or 6 weeks postsurgical bilateral oophorectomy with or without hysterectomy
   * or of childbearing potential, has a negative serum pregnancy test at screening and prior to start the study drug in each period, and abstain from sexual intercourse or agrees to using effective contraceptive methods (e.g., intrauterine device, hormonal contraceptive drug, tubal ligation or female barrier method with spermicide) during the study until completion of the follow-up procedures
4. A male is eligible to enter and participate in this study if he: agrees to abstain from sexual intercourse with females of childbearing potential or lactating females; or is willing to use a condom/spermicide, during the study until completion of the follow-up procedures.
5. Normal electrocardiogram (ECG) with QTc <450 msec.
6. Willingness and ability to comply with the study protocol for the duration of the trial.

Exclusion Criteria:

1. Females who are pregnant, trying to get pregnant, or are lactating.
2. The subject has evidence of active substance abuse that may compromise safety, pharmacokinetics, or ability to adhere with protocol instructions.
3. A positive pre-study hepatitis B surface antigen, positive hepatitis C antibody, or positive human immunodeficiency virus-1 (HIV-1) antibody result at screening.
4. Subjects with a personal history of cardiac disease, symptomatic or asymptomatic arrhythmias, syncopal episodes, or additional risk factors for torsades de pointes (heart failure, hypokalemia) or with a family history of sudden cardiac death.
5. A creatinine clearance <70 mL/min as determined by Cockcroft-Gault equation:

   CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (multiply answer by 0.85 for females) Where age is in years, weight (wt) is in kg, and serum creatinine (Scr) is in units of mg/dL [Cockcroft, 1976].
6. History of alcohol or substance abuse or dependence within 6 months of the study.
7. Use of prescription or non-prescription drugs except paracetamol at doses of up to 2 grams/day, including vitamins, herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 times the drug half-life (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise subject safety; the investigator will take advice from the manufacturer representative as necessary.
8. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days or 5 x half-life, or twice the duration of the biological effect of any drug (whichever is longer) prior to the first dose of study medication.
9. The subject is unwilling to abstain from ingesting alcohol within 48 hours prior to the first dose of study medication until collection of the final pharmacokinetic sample during each regimen.
10. Subjects who have donated blood to the extent that participation in the study would result in more than 300 mL blood donated within a 30-day period. Note: This does not include plasma donation.
11. Subjects who have a history of allergy to the study drug or drugs of this class, or a history of drug or other allergy that, in the opinion of the investigator, contraindicates participation in the trial. In addition, if heparin is used during pharmacokinetic sampling, subjects with a history of sensitivity to heparin or heparin-induced thrombocytopenia should not be enrolled.
12. Lack of suitability for participation in this study, including but not limited to, unstable medical conditions, systemic disease manifested by tendency to granulocytopenia e.g. rheumatoid arthritis and lupus erythematosus that in the opinion of the investigator would compromise their participation in the trial.
13. AST or ALT >1.5 upper limit of normal (ULN)
14. Subjects with history of renal disease, hepatic disease, and/or cholecystectomy
15. G6PD deficient
16. Abnormal methemoglobin level (more than 3 mg/dL).
17. History of antimalarial drugs use including but not limited to mefloquine, chloroquine, primaquine, artesunate, piperaquine and pyronaridine treatment within 6 months.
18. Subject who received quinacrine in last 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2016-11-18 (Actual); Primary Completion 2019-03 (Actual); Study Completion 2019-03 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve (AUC (0-∞) | 1 year
  for artemether, lumefantrine, amodiaquine and primaquine and their metabolites when given alone and in combination.
Area under the concentration-time curve AUC (0-last) | 1 year
  for artemether, lumefantrine, amodiaquine and primaquine and their metabolites when given alone and in combination.
Maximal concentration (Cmax) | 1 year
  for artemether, lumefantrine, amodiaquine and primaquine and their metabolites when given alone and in combination.

SECONDARY OUTCOMES:
Elimination clearance (CL/F) | 1 year
  of artemether, lumefantrine, amodiaquine and primaquine and their metabolites when given alone and in combination.
Terminal elimination half-life (t1/2) | 1 year
  of artemether, lumefantrine, amodiaquine and primaquine and their metabolites when given alone and in combination.
Apparent volume of distribution (Vd) | 1 year
  of artemether, lumefantrine, amodiaquine and primaquine and their metabolites when given alone and in combination.
Number of adverse events | 1 year
  Safety and tolerability parameters including adverse events, electrocardiographic changes, vital signs and biochemical assessments.
Number of event concerning of abnormal electrocardiographic | 1 year
  Safety and tolerability parameters including adverse events, electrocardiographic changes, vital signs and biochemical assessments.
Number of event concerning of abnormal vital signs | 1 year
  Safety and tolerability parameters including adverse events, electrocardiographic changes, vital signs and biochemical assessments.
Number of event concerning of abnormal laboratory values | 1 year
  Safety and tolerability parameters including adverse events, electrocardiographic changes, vital signs and biochemical assessments.
Identify polymorphisms of cytochrome 450 | 1 year
  To identify polymorphisms of cytochrome 450 related to drug metabolism from individual subject.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Tropical Medicine, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes